CLINICAL TRIAL: NCT02650869
Title: Role of Probiotics for Prevention of Necrotizing Enterocolitis in Preterm Very Low Birth Weight Infants: A Double Blind Randomized Controlled Trial
Brief Title: Role of Probiotics for Prevention of NEC in Preterm VLBW Infants
Acronym: Probiotics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sylhet M.A.G.Osmani Medical College (Other)
Responsible Party: Principal Investigator, Dr. Fazle Rabbi Chowdhury, Consultant, Sylhet M.A.G.Osmani Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SylhetMAG
Record Dates: First submitted 2015-12-31; First posted 2016-01-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Necrotizing Enterocolitis
Keywords: Necrotizing Enterocolitis; probiotics; very low birth weight
MeSH Terms: conditions — Enterocolitis, Necrotizing | interventions — Probiotics; Milk, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard care + Breast milk+ Probiotics (Experimental): The study group will be fed with probiotics at a dose of 3x109 CFU/day. (Cap TS6 probiotic + contain Bifidobacterium spp., Lactobacillus at 6x109 CFU = 6 billion CFU) dissolved with 6 ml of milk then give 3 ml (3 billion probiotics) once daily with breast milk from first feeding.
  Interventions: Dietary Supplement: Probiotics
- Standard care (Active Comparator): The control group will be given standard care without the addition of probiotics
  Interventions: Dietary Supplement: Breast milk

INTERVENTIONS:
Dietary Supplement: Probiotics — probiotics at a dose of 3x109 CFU/day. (Cap TS6 probiotic + contain Bifidobacterium spp., Lactobacillus at 6x109 CFU = 6 billion CFU manufactured by TENSALL BIO-TECH CO.LTD.Taiwan, distributed by Century Health Care, Bangladesh)
  Other Names: TS 6 Probiotics
  Arms: Standard care + Breast milk+ Probiotics
Dietary Supplement: Breast milk — Normal breast milk will be given as part of standard care
  Arms: Standard care

SUMMARY:
This prospective randomized double-blind control trial is carrying out in the neonatal unit of Sylhet MAG Osmani Medical College Hospital, Sylhet between July 2012 to December 2015 with the diagnosis of preterm (<33 weeks gestation) VLBW (birth weight <1500g) and fulfilling the inclusion criteria (able to tolerate oral feed and survive beyond 48h of life) were included in this study. Babies with suspicion of clinical sepsis, presence of perinatal asphyxia, major congenital anomaly and babies who expired due to other neonatal illness were excluded. Gestation was assessed from history of last menstrual period and after birth by new Ballard scores. A study protocol was approved by the Institutional Ethics Committee of Sylhet M.A.G Osmani Medical College, Sylhet.

DETAILED DESCRIPTION:
Background: Necrotizing enterocolitis (NEC) is the most common acquired disease of the gastrointestinal tract in preterm very low birth weight infants and associated with increased morbidity and mortality. Prophylactic enteral probiotic supplementation may play a role in reducing NEC and potentially provide benefits to preterm very low birth weight neonates. The objective was to evaluate the efficacy of orally administered probiotics in preventing necrotizing enterocolitis (NEC) in preterm very low birth weight (VLBW) infants.

This prospective, randomized double blind controlled trial is undergoing in 102 preterm (28-33 weeks gestation) VLBW (birth weight 1000-1499g) neonates fulfilling the inclusion criteria. The study group was fed with probiotics once daily with breast milk from first feeding and the control group only breast milk without the addition of probiotics. The primary outcome was the development of NEC (stage II and III). NEC is categorized by modified Bell's classification.

Probiotic supplementation reduces the frequency of necrotising enterocolitis in preterm neonates with very low birth weight. It is also associated with faster achievement of full enteral feeding and shorter duration of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* All newborn infant preterm (<33 weeks gestation to 28 weeks gestation) VLBW (birth weight <1500gm to 1000 gm)
* Able to tolerate oral feed
* Informed consent by the parents or guardian

Exclusion Criteria:

* Evidence or suspicion of clinical sepsis before the baby is randomised
* Presence of perinatal asphyxia
* Presence of major congenital anomali
* Death within first week of life due to other neonatal illness

Ages: 1 Week to 33 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2012-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Necrotizing Enterocolitis: Occurrence of NEC (stage II and III) by Modified Bell's classification | 10 days
  The occurrence of NEC (stage II and III) by modified Bell's classification

SECONDARY OUTCOMES:
Enteral feeding | 10 days
  days to achieve full enteral feeding
Hospital stay | 10 days
  maximum days of hospital stay
weight in Kg | 10 days
  weight in kg

CONTACTS AND LOCATIONS:
Overall Officials: Prof. M. Monojjir Ali, FCPS, Study Chair — Professor and Head, Department of Paediatrics, Sylhet M.A.G.Osmani Medical College

REFERENCES:
- [Background] Sharma R, Tepas JJ 3rd, Hudak ML, Mollitt DL, Wludyka PS, Teng RJ, Premachandra BR. Neonatal gut barrier and multiple organ failure: role of endotoxin and proinflammatory cytokines in sepsis and necrotizing enterocolitis. J Pediatr Surg. 2007 Mar;42(3):454-61. doi: 10.1016/j.jpedsurg.2006.10.038. PMID 17336180
- [Background] Forchielli ML, Walker WA. The effect of protective nutrients on mucosal defense in the immature intestine. Acta Paediatr Suppl. 2005 Oct;94(449):74-83. doi: 10.1111/j.1651-2227.2005.tb02159.x. PMID 16214770
- [Background] Neish AS, Gewirtz AT, Zeng H, Young AN, Hobert ME, Karmali V, Rao AS, Madara JL. Prokaryotic regulation of epithelial responses by inhibition of IkappaB-alpha ubiquitination. Science. 2000 Sep 1;289(5484):1560-3. doi: 10.1126/science.289.5484.1560. PMID 10968793
- [Background] Deshpande G, Rao S, Patole S. Probiotics for prevention of necrotising enterocolitis in preterm neonates with very low birthweight: a systematic review of randomised controlled trials. Lancet. 2007 May 12;369(9573):1614-20. doi: 10.1016/S0140-6736(07)60748-X. PMID 17499603